CLINICAL TRIAL: NCT02871804
Title: Comparison of Resection During Distal Pancreatectomy of the Splenic Vein Either Together With the Pancreatic Parenchyma or After Isolation: A Multicentre, Prospective, Randomized Phase III Trial
Brief Title: Combined Resection vs. Separated Resection After Mobilization of Splenic Vein During Distal Pancreatectomy
Acronym: COSMOS-DP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Hiroki Yamaue, Professor, Wakayama Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COSMOS-DP trial
Record Dates: First submitted 2016-07-27; First posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- separated resection of the splenic vein (Active Comparator): separated resection of the splenic vein from the pancreatic parenchyma before ligation and division during distal pancreatectomy using mechanical staplers.
  Interventions: Procedure: separated resection of the splenic vein
- combined resection of the splenic vein (Experimental): combined resection of the splenic vein with the pancreatic parenchyma before ligation and division during distal pancreatectomy using mechanical staplers.
  Interventions: Procedure: combined resection of the splenic vein

INTERVENTIONS:
Procedure: combined resection of the splenic vein — combined resection of the splenic vein with the pancreatic parenchyma before ligation and division during distal pancreatectomy using mechanical staplers.
  Arms: combined resection of the splenic vein
Procedure: separated resection of the splenic vein — separated resection of the splenic vein from the pancreatic parenchyma before ligation and division during distal pancreatectomy using mechanical staplers.
  Arms: separated resection of the splenic vein

SUMMARY:
Eligible patients will be centrally randomized to either Arm A (resection of the splenic vein after isolation from the pancreatic parenchyma) or Arm B (co-resection of the vein together with the pancreas).

DETAILED DESCRIPTION:
In distal pancreatectomy, it is customary to ligate and divide the splenic vein after isolating it from the pancreatic parenchyma. This is considered essential to prevent disruption of the stump of the splenic vein and the consequent intra-abdominal haemorrhage in the event of pancreatic fistula. This procedure can be technically demanding, especially when the vein is firmly embedded in the pancreatic parenchyma. The objective of this trial is to confirm the non-inferiority of resection of the splenic vein embedded in the pancreatic parenchyma compared with the conventional technique of isolating the splenic vein before resection during distal pancreatectomy using a mechanical stapler.

ELIGIBILITY:
Inclusion Criteria:

* Elective open or laparoscopic distal pancreatectomy for diseases of the pancreatic body and tail
* ECOG Performance Status (PS) = 0-1
* Age ≥ 20 years old
* Maintenance of functioning of the major organs (bone marrow, liver, kidney, lung, etc.) (a) White blood cells ≥ 2,500/mm3 (b) Haemoglobin ≥ 9.0 g/dL (c) platelets ≥ 100,000/mm3 (d) Total bilirubin ≤ 2.0 mg/dL (e) Creatinine ≤ 2.0 mg/dL (v) Sufficient judgement to understand the study and to provide written informed consent

Exclusion Criteria:

* Splenic vein-preserving distal pancreatectomy
* Superior mesenteric vein or portal vein invasion
* Pancreatic trauma
* Preoperative inflammatory pancreatic disease (pancreatitis)
* Requirement of anti-coagulant treatment during or after surgery. Anti-coagulant treatment at 24 hrs after surgery is allowed.
* Severe ischemic cardiovascular disease
* Liver cirrhosis or active hepatitis
* Need for oxygen due to interstitial pneumonia or lung fibrosis
* Dialysis due to chronic renal failure
* Need for surrounding organ resection (stomach, colon, etc.), excluding the left adrenal gland and gall bladder
* Active multiple cancer that is thought to influence the occurrence of adverse events
* Difficulty with study participation due to psychotic disease or symptoms
* Inappropriate use of the stapler
* Inappropriate for the study objectives

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-08 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
the incidence of pancreatic fsitula grade B/C | 6 months after operation

SECONDARY OUTCOMES:
the incidence of pancreatic fsitula of all grades | 6 months after operation
the incidence of pancreatic fsitula grade C | 6 months after operation
the incidenceof intra-abdominal haemorrhage | 6 months after operation
the incidence of all complications | 6 months after operation
comparison of the thickness of the resected pancreatic parenchyma with the incidence of PF grade B/C | 6 months after operation
mortality | 6 months after operation
the incidence of thrombosis of the splenic vein | 6 months after operation
the operative time | during operation
volume of blood loss | during operation
thickness of the resected pancreatic parenchyma | during operation
haemostasis of the staple line | during operation
integrity of the staple line | during operation
the incidence of pancreatic injury | during operation
need for additional sutures to securely close the pancreatic stump | during operation
time needed for pancreatic transection | during operation
duration of drainage tube placement | 6 months after operation
postoperative hospital stay duration | 6 months after operation
the incidence of conversion from laparoscopic surgery to open surgery | during operation

CONTACTS AND LOCATIONS:
Overall Officials: Hiroki Yamaue, MD, PhD, Principal Investigator — Wakayama Medical University
Locations (1):
- Wakayama Medical University, Wakayama, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yamada S, Fujii T, Sonohara F, Kawai M, Shibuya K, Matsumoto I, Fukuzawa K, Baba H, Aoki T, Unno M, Satoi S, Kishi Y, Hatano E, Uemura K, Horiguchi A, Sho M, Takeda Y, Shimokawa T, Kodera Y, Yamaue H. Safety of Combined Division vs Separate Division of the Splenic Vein in Patients Undergoing Distal Pancreatectomy: A Noninferiority Randomized Clinical Trial. JAMA Surg. 2021 May 1;156(5):418-428. doi: 10.1001/jamasurg.2021.0108. PMID 33656542
- [Derived] Yamada S, Fujii T, Kawai M, Shimokawa T, Nakamura M, Murakami Y, Satoi S, Eguchi H, Nagakawa Y, Kodera Y, Yamaue H. Splenic vein resection together with the pancreatic parenchyma versus separated resection after isolation of the parenchyma during distal pancreatectomy (COSMOS-DP trial): study protocol for a randomised controlled trial. Trials. 2018 Jul 11;19(1):369. doi: 10.1186/s13063-018-2756-7. PMID 29996884